CLINICAL TRIAL: NCT02182895
Title: Safety and Efficacy of Saxagliptin for Glycemic Control in Non-Critically Ill Hospitalized Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rajesh K. Garg, Rajesh Garg, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001095
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin group (Experimental): DPP4 inhibitor therapy group will receive saxagliptin 2.5 to 5 mg daily in addition to correctional sliding scale insulin therapy before each meal and bedtime.
  Interventions: Drug: Saxagliptin
- Standard therapy group (No Intervention): Standard therapy group will receive basal-bolus insulin starting at a dose of 0.5 units/kg/day; given half as insulin glargine and half as insulin aspart. In addition, the standard therapy group will receive the correctional sliding scale insulin therapy before each meal and bedtime.

INTERVENTIONS:
Drug: Saxagliptin — 2.5-5 mg daily
  Other Names: Onglyza; DPP4 inhibitor
  Arms: Saxagliptin group

SUMMARY:
The purpose of this research study is to test the safety and efficacy of a drug called saxagliptin (Onglyza) for treatment of type 2 diabetes in non-critically ill hospitalized patients who have an HbA1c of 7.5 or lower, on 1 or no non-insulin agent at home, or an HbA1c ≤7.0% on ≤ 2 non-insulin agents at home.

DETAILED DESCRIPTION:
The current professional organization guidelines recommend insulin as the preferred treatment for hospitalized patients. It is recommended that most critically ill patients should receive insulin infusion therapy and non-critically ill patients should receive basal bolus insulin therapy in the hospital.

The study will test the hypothesis that treatment with saxagliptin is non-inferior to treatment with basal bolus insulin in this group of patients during their hospital stay. The study will evaluate the effect of saxagliptin, a DPP4 inhibitor, on glycemic control in non-critically ill hospitalized patients with type 2 diabetes mellitus (T2DM)

The primary outcome will be mean daily blood glucose levels during hospital days 2 to 5. The study is designed to detect a non-inferiority margin of 20% in the saxagliptin group as compared to the control group

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM and HbA1C ≤7.5% on ≤1 non-insulin hypoglycemic agent or HbA1C ≤7.0% on ≤2 non-insulin hypoglycemic agents admitted to the hospital for a non-critical illness.
* Written informed consent.

Exclusion Criteria:

* Admitted to or expected to require admission to ICU
* Patients with a history of diabetic ketoacidosis or hyperosmolar state
* HbA1c >7.5% at the time of admission or within 3 months before admission
* Insulin requiring before admission
* Unable to take oral food or medications
* Systemic steroid use
* Pregnancy or breastfeeding
* Women of Child-Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and up to 4 weeks after the last dose of study drug.
* History of pancreatitis or active gallbladder disease
* End stage renal disease on dialysis
* Hypersensitivity to saxagliptin or another contraindication to DPP4 inhibitors
* Subject unable to give informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh K Garg, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.

REFERENCES:
- [Derived] Garg R, Schuman B, Hurwitz S, Metzger C, Bhandari S. Safety and efficacy of saxagliptin for glycemic control in non-critically ill hospitalized patients. BMJ Open Diabetes Res Care. 2017 Mar 29;5(1):e000394. doi: 10.1136/bmjdrc-2017-000394. eCollection 2017. PMID 28405346

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin Group: saxagliptin 2.5-5 mg daily
- Standard Therapy Group: No saxagliptin treatment
Period: Overall Study
Arm/Group | Saxagliptin Group | Standard Therapy Group
Started | 35 | 37
Completed | 33 | 33
Not Completed | 2 | 4
Not completed — Discharged from hospital within 24 hours | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin Group | Standard Therapy Group | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 67 (10) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 13 | 17 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 26 | 30 | 56
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (12.2) | 32.6 (6.5) | 33.6 (10)

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose Levels During Hospital
Description: mean of average daily blood blood glucose for each patient day
Time Frame: Hospital days 2-5
Population: Inpatients with diabetes
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
mg/dL | 154.8 (28.2) | 156.0 (32.1)

2. Secondary Outcome: Percentage of Blood Glucose Readings in 70-140 mg/dL Range
Description: Percentage of BG readings in the desired range of 70-140 mg/dl out of all avaialble BG readings.
Time Frame: Days 2 to 5
Population: completed subjects
Measure: Number; unit: % of blood glucose readings
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
% of blood glucose readings | 42 | 37

3. Secondary Outcome: Dose of Insulin
Description: Average daily amount of insulin used
Time Frame: Days 2 to 5
Population: completed subjects
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
Units | 2.4 (3.3) | 13.3 (12.9)

4. Secondary Outcome: Incidence of Hypoglycemia (BG <70 mg/dL)
Description: Number of BG readings <70 mg/dL in each group
Time Frame: Days 2 to 5
Population: completed
Measure: Number; unit: number of events
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
number of events | 1 | 1

5. Secondary Outcome: Incidence of Hyperglycemia (Blood Glucose >200 mg/dL)
Description: Proportion of BG readings in the severe hyperglycemic range.
Time Frame: Days 2 to 5
Population: completed
Measure: Number; unit: % of blood glucose readings >200
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
% of blood glucose readings >200 | 6 | 10

6. Secondary Outcome: Variability in Glucose Levels
Description: Mean amplitude of glycemic excursions
Time Frame: Days 2 to 5
Population: Patients who allowed a CGMS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 20 | 16
mmol/L | 2.72 (1.60) | 3.93 (2.03)

7. Secondary Outcome: Length of Hospital Stay
Description: Number of days in hospital
Time Frame: Admission to discharge, an expected average of 5 days
Population: completed
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
days | 8.0 (14.6) | 6.4 (5.4)

8. Secondary Outcome: Patient Satisfaction
Description: Diabetes Treatment Satisfaction Questionnaire - InPatient (DTSQ-IP). This questionnaire had 14 items that were scored on a scale of 0 to 6. Total score for each subjects could range from 0-84. Higher score means better satisfaction.
Time Frame: At the time of discharge or Day 5
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Saxagliptin Group | Standard Therapy Group
Number analyzed (Participants) | 33 | 33
Score | 70 (12) | 75 (11)

ADVERSE EVENTS:
Time Frame: During the study period.
Arm/Group | Saxagliptin Group | Standard Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saxagliptin Group (N=33) | Standard Therapy Group (N=33)
Failure to control hyperglucycemia (Endocrine disorders) | 2 (2) | 0 (0) — Study drug stopped

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No